CLINICAL TRIAL: NCT07226882
Title: A PHASE 3, PLACEBO-CONTROLLED, DOUBLE-BLINDED, RANDOMIZED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF DIFFERENT VACCINATION SCHEDULES OF 6-VALENT OSPA-BASED LYME DISEASE VACCINE, VLA15, IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn About Different Dosing Schedules of a Lyme Disease Vaccine in Healthy Adults
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C4601019
Record Dates: First submitted 2025-10-13; First posted 2025-11-12 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Lyme Borreliosis
Keywords: Lyme disease; Lyme Borreliosis, Nervous System; Lyme; Lyme Disease Vaccine
MeSH Terms: conditions — Lyme Disease; Lyme Neuroborreliosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Third-party unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Participants will receive 4 doses of VLA15 and 1 dose of placebo injection at different visits. Placebo will be given at Visit 3. Injections will be given as intramuscular shots.
  Interventions: Biological: VLA15; Biological: Placebo
- Group 2 (Experimental): Participants will receive 4 doses of VLA15 and 1 dose of placebo injection at different visits. Placebo will be given at Visit 5. Injections will be given as intramuscular shots.
  Interventions: Biological: VLA15; Biological: Placebo
- Group 3 (Experimental): Participants will receive 4 doses of VLA15 and 1 dose of placebo injection at different visits. Placebo will be given at Visit 7. Injections will be given as intramuscular shots.
  Interventions: Biological: VLA15; Biological: Placebo
- Group 4 (Experimental): Participants will receive 4 doses of VLA15 and 1 dose of placebo injection at different visits. Placebo will be given at Visit 9. Injections will be given as intramuscular shots.
  Interventions: Biological: VLA15; Biological: Placebo

INTERVENTIONS:
Biological: VLA15 — Participants will receive IM injection of 6-valent OspA-based Lyme disease vaccine
Biological: Placebo — Saline

SUMMARY:
The purpose of this study is to learn about the safety and effects of the Lyme disease vaccine (called VLA15) when given at different time points.

This study is seeking participants who:

* are generally healthy and between 18 and 44 years of age,
* have never had a vaccine for Lyme disease before,
* are not currently taking, or haven't recently taken, medicines like chemotherapy, blood products, or blood thinners, and
* are not pregnant or breastfeeding and do not plan to become pregnant while receiving the study vaccine.

All participants in this study will receive a total of 5 doses through a shot in the upper arm. Four doses will be the study vaccine (VLA15), and 1 dose will be saltwater.

The study will compare the experiences of people receiving the study vaccine at different time points. This will help see if the study vaccine is safe and will help understand its effect on the body.

Participants will take part in this study for about 2 years. During this time, the participants will have 11 planned visits - 8 will be at the study clinic and 3 will be done over the phone. The clinic visits may include having a health check, giving a small amount of blood (about 20 mL or 4 teaspoons), and getting the study vaccine or saltwater as a shot.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, parallel-group, placebo-controlled, double-blinded (third-party unblinded) study to evaluate the safety, tolerability, and immunogenicity of different vaccination schedules of the 6-valent OspA-based Lyme disease (LD) vaccine, VLA15, in healthy participants 18 through 44 years of age.

Participants will be randomized in a 1:1:1:1 ratio to 1 of the 4 parallel study groups. Each participant will receive 4 doses of VLA15 and 1 dose of placebo (saline) at different time points. This study will use an external data monitoring committee (EDMC). The EDMC is independent of the Pfizer study team and includes only external members. The EDMC charter describes the role of the EDMC in more detail.

Approximately 200 participants will be enrolled in the study.

Healthy individuals 18 through 44 years of age who are willing to comply with all study procedures and provide signed informed consent will be enrolled. Pregnant or breastfeeding individuals and fertile individuals who are unwilling or unable to use effective contraceptive methods as outlined in this protocol will not be enrolled. Individuals who have contraindication to vaccination, conditions or treatments that can inhibit the ability to mount an immune response to a vaccine, or other conditions that may increase the risk of study participation will be excluded from this study. Individuals who have previously received a licensed or investigational vaccine for LD will also be excluded from this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are healthy as determined by medical history and clinical judgment.
* Participants willing and able to comply with all scheduled visits, IP receipt, and other procedures throughout the study.
* Able to provide Informed Consent.

Exclusion Criteria:

* Pregnant or breastfeeding participants.
* Allergies or contraindications to vaccines or their components.
* Health issues including: blood clotting deficiencies, immunodeficiencies, bone marrow disorder, or uncontrolled psychiatric conditions.
* Receipt of therapies to treat malignancies, blood/plasma products and immunoglobulins, systemic corticosteroids and immunosuppressants, or anticoagulant therapy in recent medical history.
* Any prior Lyme disease vaccination, or recent or concurrent participation in a separate interventional study.
* Staff or direct family of the study site staff and Sponsor.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2028-02-14 (Estimated); Study Completion 2028-02-14 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Concentration (GMC) of Anti-Outer Surface Protein A (OspA) Immunoglobulin G (IgG) | At 1 month after the fourth VLA15 dose
Geometric Mean Fold Rise (GMFR) of Anti-Outer Surface Protein A (OspA) Immunoglobulin G (IgG) Concentrations | Before the first dose to 1 month after the fourth VLA15 dose
Percentage of Participants With Local Reactions For Each Group | Within 7 days after each vaccination
Percentage of Participants With Systemic Events For Each Group | Within 7 days after each vaccination
Percentage of Participants With Adverse Events (AEs) For Each Group | Within 1 month after each vaccination
Percentage of Participants With Serious Adverse Events (SAEs) For Each Group | From the time the participant provides informed consent up to approximately 6 months after the last vaccination
Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) For Each Group | From the time the participant provides informed consent up to approximately 6 months after the last vaccination

SECONDARY OUTCOMES:
Geometric Mean Concentration (GMC) of Anti-Outer Surface Protein A (OspA) Immunoglobulin G (IgG) | At 1 month after the third VLA15 dose
Geometric Mean Fold Rise (GMFR) of Anti-Outer Surface Protein A (OspA) Immunoglobulin G (IgG) Concentrations | Before the first dose to 1 month after the third VLA15 dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Preferred Primary Care Physicians, Preferred Clinical Research (Ofc 18), Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research-St. Clair, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Amherst Family Practice, P.C., Winchester, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4601019